CLINICAL TRIAL: NCT05584722
Title: Risk and Resilience in Pulmonary Arterial Hypertension and Genetically Susceptible Individuals
Acronym: RARE-PAH
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Anna Hemnes, MD, Vanderbilt University Medical Center
Other Study IDs: 221437; 1R01FD007627 (FDA)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension; Unaffected Mutation Carriers: Healthy Participants With a Known BMPR2 Gene Mutation and Normal Pulmonary Pressure and RV Function on Echo; Healthy Individuals With no Cardiopulmonary Disease
Keywords: pulmonary hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We plan to collect the following samples on selected subjects:
  DNA, RNA, serum, and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic or Heritable Pulmonary Arterial Hypertension: Patients diagnosed with pulmonary arterial hypertension, either idiopathic or heritable, defined according to standard criteria.
- Unaffected Mutation Carriers: Healthy participants with a known BMPR2 gene mutation and normal pulmonary pressure and RV function on echo.
- Healthy Controls: Healthy individuals without cardiopulmonary disease

SUMMARY:
Pulmonary arterial hypertension (PAH) is a severe disease with a delayed diagnosis and markedly elevated mortality. High-risk populations, such as those with known genetic defects, provide a unique opportunity to determine the features of susceptibility and resilience to PAH. This proposal will fundamentally overturn the prevailing understanding of PAH by creating molecularly-driven signatures of susceptibility and resilience, provide novel insight into disease severity, and potentially identify new therapeutic targets.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is an orphan disease with a delayed diagnosis and markedly elevated mortality from right heart failure. Despite nearly a dozen FDA-approved drugs for PAH, median survival is only seven years. All approved therapies target one of three vasodilatory pathways, and none are disease modifying. This study has two objectives: 1) Understand dynamic and static relationships between molecular markers and PAH progression and resilience; 2) Identify molecular features of PAH risk and resilience in individuals harboring a PAH-causing mutation. It is unknown why some at risk individuals develop PAH and others do not. BMPR2 mutations are present in about 30% of patients with PAH but clinical penetrance is only 20%. Unaffected BMPR2 mutation carriers (UMCs) are a unique and understudied population that may also provide clues to disease trajectory in patients with clinical PAH. Longitudinal natural history studies with molecular profiling in PAH are lacking. Most molecular profiling studies in PAH are cross-sectional which limits understanding of how disease progression and disease markers relate over time. The Investigators propose a strategy of dense clinical and molecular phenotyping at multiple timepoints to overcome inferential limitations of cross-sectional studies. This application will leverage the clinical and research infrastructure built at Vanderbilt over the past 35 years in our study of PAH patients. The investigators share an extensive published record of recruiting patients with this rare disease and related UMCs. The Investigators hypothesize that a comprehensive understanding of risk and resilience over time in patients and genetically susceptible individuals will provide insight into disease severity and identify novel therapeutic targets in patients with PAH. Aim 1 will identify static and dynamic molecular features of disease progression and resilience. 1a: Perform serial clinical, proteomic, and gene expression profiling in HPAH, IPAH, and healthy controls 3 times over 4 years. Bioinformatic and network medicine analyses will identify proteins and RNAs associated with changes in clinical outcomes, functional capacity, and RV function in the parent cohort and two external validation cohorts.1b: Test whether adding molecular risk/resilience markers will improve the performance of a widely used PAH risk prediction tool (REVEAL 2.0 Risk Score). Aim 2 will identify the clinical and molecular factors that promote resilience and susceptibility to PAH in a longitudinal cohort of UMCs. UMCs will undergo serial clinical and molecular phenotyping as in Aim 1. Proteins/genes that mirror PAH are "risk factors" and those that mirror a healthy population are "resilience factors". Explanatory models will be developed and tested in validation cohorts. The Investigators will test UMC risk and resilience features for associations with clinical outcomes in PAH patients and risk prediction performance. These studies will identify signatures of risk and resilience to PAH progression and penetrance, offering an initial step toward personalizing care and surveillance guided by biologic data.

ELIGIBILITY:
Inclusion Criteria:

* Children and Adults, aged 15 - 80
* Diagnosed with idiopathic or heritable, pulmonary arterial hypertension (PAH), defined according to standard criteria
* Unaffected Mutation Carriers: Healthy participants with a known BMPR2 gene mutation and normal pulmonary pressure and RV function on echo
* Healthy Controls: Healthy individuals without cardiopulmonary disease.
* WHO functional class I-III
* Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included. Adjustments in IV prostacyclin for side effect management are allowed.

Exclusion Criteria:

* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition that limits activity.
* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable
* Functional class IV heart failure
* Requirement of > 2 diuretic adjustment in the prior three months.

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Diagnosed with idiopathic or heritable, pulmonary arterial hypertension (PAH), defined according to standard criteria
  * Unaffected Mutation Carriers: Healthy participants with a known BMPR2 gene mutation and normal pulmonary pressure and RV function on echo
  * Healthy Controls: Healthy individuals without cardiopulmonary disease.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by the emPHasis-10 | Baseline to 32 months
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items that address breathlessness, fatigue, control, and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Change in Quality of Life as measured by the Pediatric Quality of Life Inventory Version 4.0 | Baseline to 32 months
  The PedsQL (Pediatric Quality of Life Inventory) is a modular instrument for measuring health-related quality of life in children and adolescents ages 2 to 18. The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure that consists of 23 items applicable for healthy school and community populations, as well as pediatric populations with acute and chronic health conditions.
Change in meters walked in six-minute walk distance (meters) | Baseline to 32 months
  The 6MWT measures the distance (in meters), a participant can walk at a comfortable speed on a flat, hard surface in 6 minutes. The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out daily physical activities.
Change in diffusing capacity for carbon monoxide (DLCO) on the Pulmonary Function Test | Baseline to 32 months
  Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange.
  DLCO measures the quantity of carbon monoxide (CO) transferred per minute from alveolar gas to red blood cells in pulmonary capillaries and is expressed as mL/min/mm Hg.
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE), expressed in mm. | Baseline to 32 months
  Change from baseline in Tricuspid Annular Plane systolic Excursion (TAPSE) expressed in mm on echocardiogram results at 12-16 months and 24-32 months.
Change in Tricuspid Annular Velocity (S'), as assessed by echocardiogram results, expressed in cm/sec | Baseline to 32 months
  Change from baseline in Tricuspid Annular Velocity (S') on echocardiogram results at 12-16 months and 24-32 months and expressed in cm/sec.
Change in Estimated Right Ventricle (RV) Systolic Pressure, as assessed by echocardiogram results, expressed in mmHg | Baseline to 32 months
  Change from baseline in the estimated right ventricular systolic pressure on echocardiogram results at 12-16 months and 24-32 months and expressed in mmHg.
Change in Right Ventricle (RV) Free Wall Longitudinal Strain, as assessed by echocardiogram results, and expressed as percent (%) change in myocardial deformation. | Baseline to 32 months
  Change from baseline in right ventricle free wall longitudinal strain on echocardiogram results at 12-16 months and 24-32 months and expressed as percent (%) change in myocardial deformation.
Change in Daily Step Count as measured by the mHealth device mean daily step count | Baseline to 32 months
  Change from the baseline activity monitoring period to the 12-16 month activity monitoring period to the 24-32 month activity monitoring period. Data obtained by the mHealth device.
Change in Resting Heart Rate (beats per minute) | Baseline to 32 months
  Monitored regularly using activity tracking device (per second when active, per 5 seconds when inactive). Subject's resting and peak exercise heart rate will also be recorded at baseline, 12-16 months, and 24-32 months. Targets exercise capacity. Heart rate is expressed as beats per minute.
Intensity of activity | Baseline to 32 months
  Intensity of activity is categorized as rest, light, moderate, and vigorous based on calculated metabolic equivalents.
Number of patients with a PAH-related Hospitalization Incidence | Baseline to 32 months
  To assess PAH-related hospitalization incidences from baseline to 12-16 months and 24-32 months. Number of patients will be assessed.
Change in Patient Medication Regimen, as measured by percentage (%) of subjects with a change in medication regimen | Baseline to 32 months
  Change from baseline in patient medication regimen from baseline to 12-16 months and 24-32 months as measured by percentage (%) of subjects with a change in medication regimen.
Number of patients with an incidence of death | Baseline to 32 months
  To assess incidences of death from baseline to 12-16 months and 24-32 months. Number of patients will be assessed.
Number of patients with an incidence of lung transplantation | Baseline to 32 months
  To assess incidences of lung transplantation from baseline to 12-16 months and 24-32 months. Number of patients will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, Principal Investigator — Vanderbilt Medical Center; Anna Hemnes, MD, Principal Investigator — Vanderbilt Medical Center; Eric Austin, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No